CLINICAL TRIAL: NCT02489071
Title: Cognitive Intervention After a Brain Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-7277-CE
Record Dates: First submitted 2015-06-16; First posted 2015-07-02 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brain Training (Experimental): 8-session cognitive training program
  Interventions: Behavioral: Brain Training Program
- Brain Health (Experimental): 8-session cognitive education program
  Interventions: Behavioral: Brain Health Program
- Control (No Intervention): Wait-list control group

INTERVENTIONS:
Behavioral: Brain Training Program
  Arms: Brain Training
Behavioral: Brain Health Program
  Arms: Brain Health

SUMMARY:
This study evaluates the feasibility and utility of two behavioural programs designed to reduce cognitive impairments secondary to brain tumors and/or their treatment. One-third of participants will complete training in either program, with the remaining third a wait-list control group.

DETAILED DESCRIPTION:
Cognitive impairments (including problems with attention, memory or executive functions) are common in people with brain tumors, as a result of the disease and/or treatment effects. These deficits, even when relatively mild, can interfere with interpersonal relationships, occupational activities, functional independence, and quality of life. They may also contribute to caregiver burden.

Building on research in other cognitively-impaired populations, in this study we compare two behavioural interventions. The Brain Training (BT) and Brain Health (BH) interventions each offer a structured yet client-centered program through 8 weekly individual treatment sessions and between-session exercises. Contents include mindfulness practice, strategy training, and supportive psychoeducation including counseling around lifestyle factors to promote brain functioning.

Using a prospective randomized controlled design, 54 brain tumor patients are being enrolled in one of three study arms: BT, BH, or standard care (wait-list control). A battery of outcome measures is being administered (1) prior to intervention, (2) after the 8-week behavioural intervention (or wait-list) period, and (3) after an additional 4 months to evaluate longer-term outcomes. Analyses of variance will examine treatment effects, with regression analyses to explore moderating effects of participant demographics, severity of baseline cognitive impairment, and tumor and treatment factors (e.g., tumor location, radiation dose and distribution). Results of this trial will lay the groundwork for implementation of evidence-based supportive care to reduce and manage cognitive impairments following a brain tumor.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older
2. fluent in English
3. able to provide informed consent to all procedures
4. diagnosis of a brain tumor
5. indication of lasting post-treatment cognitive deficits (e.g., from clinical presentation, prior neuropsychological assessment, and/or self-report)
6. sufficient motor and sensory functioning to complete study activities
7. availability to complete all study activities
8. for patients treated with cranial radiation, at least 3 months post-radiation

Exclusion Criteria:

(1) comorbid neurological or psychiatric disorder or other medical condition suspected to influence cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in cognitive composite score | baseline, 2 months (0-2 weeks post-training), 6 months (4 months post-training)
  Summation of standardized change scores on neuropsychological tests

SECONDARY OUTCOMES:
Change in functional composite score | baseline, 2 months (0-2 weeks post-training), 6 months (4 months post-training)
  Summation of standardized change scores on measures of occupational functioning
Change in quality of life composite score | baseline, 2 months (0-2 weeks post-training), 6 months (4 months post-training)
  Summation of standardized change scores on measures of affect, perceived self-efficacy, and illness burden
Change in caregiver quality of life composite score | baseline, 2 months (0-2 weeks post-training), 6 months (4 months post-training)
  Summation of standardized change scores on measures of affect and caregiver burden

CONTACTS AND LOCATIONS:
Overall Officials: Kim Edelstein, PhD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Richard NM, Bernstein LJ, Mason WP, Laperriere N, Maurice C, Millar BA, Shultz DB, Berlin A, Edelstein K. Cognitive rehabilitation for executive dysfunction in brain tumor patients: a pilot randomized controlled trial. J Neurooncol. 2019 May;142(3):565-575. doi: 10.1007/s11060-019-03130-1. Epub 2019 Mar 7. PMID 30847839